CLINICAL TRIAL: NCT01034670
Title: Advanced Gastrointestinal Endoscopic Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in personnel and cessation of funding
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-15766; NCI-2021-03446 (Other: NCI Trial Identifier); U54CA136465 (NIH)
Record Dates: First submitted 2009-11-13; First posted 2009-12-17 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal Diseases; Gastric (Stomach) Cancer; Gastrointestinal Stromal Tumor (GIST)
MeSH Terms: conditions — Gastrointestinal Diseases; Stomach Neoplasms; Gastrointestinal Stromal Tumors | interventions — Fluorescein; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- endoscopy arm (Experimental): imaging performed in conjunction with the regularly scheduled endoscopy during which the newer imaging techniques will be used to detect premalignant conditions. includes wide field fluorescence, microscopy, Raman spectroscopy and/or ultrasound.
  Interventions: Device: Dual axis endoscopic microscope; Device: wide field fluorescence system; Device: CellVizio; Drug: fluorescent Peptide; Drug: fluorescein; Drug: indocyanine green

INTERVENTIONS:
Device: Dual axis endoscopic microscope — This is a device that is used in the accessory port of a standard endoscope and allows visualization of microscopic areas of mucosa.
  Other Names: Stanford
Device: wide field fluorescence system — This is a modification to the existing narrow band endoscope from Olympus that incorporates different filters on the source and collecting optics to enable fluorescence imaging. It is used as is a standard endoscope.
  Other Names: Olympus
Device: CellVizio — Minimicroscope--this is an FDA approved fiber-based microscope that we will use according to the manufacturers protocols.
  Other Names: Mauna Kea Technologies
Drug: fluorescent Peptide — microdosing; Topical through the endoscope
  Other Names: GMP
Drug: fluorescein — 100 mcg topical
  Other Names: fluorophore
Drug: indocyanine green — 100 mcg topical
  Other Names: ICG

SUMMARY:
To develop new methods to detect malignant and premalignant conditions of the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:patients be at least 18 years of age,

Either genders

All ethnic backgrounds will be considered.

Patients who are scheduled for endoscopy by one of the investigators will be asked if they are interested in participating in the study.

The study will be open to all patients undergoing endoscopy that do not have exclusion criteria. We will ask all patients if they are participating in any other studies. If they are participating in any other study then we will ask them for more information to determine whether there could be any harm from participating in both studies and if there is then they will not be enrolled. Exclusion Criteria:Patients with unstable vital signs will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shai Friedland, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endoscopy Arm
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Endoscopy Arm
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Imaging of the Mucosa
Description: Detection of mucosa abnormailities as a first step in the goal of detection of neoplasia
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopy Arm
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Endoscopy Arm
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT01034670/Prot_000.pdf